CLINICAL TRIAL: NCT06679426
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Study Evaluating the Safety and Efficacy of Conestat Alfa As a Treatment for Angiotensin-Converting Enzyme-Inhibitor-Induced Angioedema
Brief Title: Safety and Efficacy of Conestat Alfa for ACE-Induced Angioedema
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, Jonathan Bernstein, Adjunct Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-0561
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-07

CONDITIONS: ACE Inhibitor-Induced Angioedema
Keywords: Ruconest, conestat alpha, ACE inhibitor, angioedema, treatment, outcome, safety
MeSH Terms: conditions — Angioedema | interventions — conestat alfa

STUDY DESIGN:
Intervention Model Description: This Phase III study is designed as a randomized, double-blind, two-armed, placebo-controlled study (Figure 2). It will be conducted at two centers in the United States. The primary aim is to compare the efficacy of conestat alfa with a placebo in the treatment of ACE-I-induced AE based on the TMDC endpoint, assess its safety and tolerability, as well as compare its efficacy compared to the placebo based on the TOSR endpoint. Moreover, the proportion of patients in each arm who are hospitalized, admitted to the ICU, or who require an airway intervention will be compared.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be conducted as a double-blind, placebo-controlled trial. The appearance of the prefilled device containing placebo will be indistinguishable from those containing conestat alfa. The blinding will be maintained throughout the duration of the study for the subject. As such, only investigators and study staff blinded to the treatment assignments will be responsible for monitoring the patient and assessing efficacy and safety outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational product (Active Comparator): Human recombinant C1-INH, also known as conestat alfa (Ruconest™), has been purified from the breast milk of genetically modified rabbits. Conestat alfa targets activated C1s, kallikrein, factor XIIa, and factor XIa. Inhibition kinetics are comparable to plasma-derived human C1-INH. The elimination half-life is approximately 2.5 hours.37 One vial consists of 2100 units, which corresponds to 2100 units per 14 mL after reconstitution, resulting in a concentration of 150 units/mL. One unit of activity corresponds to C1 esterase inhibiting activity in 1 mL of normal plasma. Each vial also contains 19.5 mg of sodium.41 In order to administer 4200 IU of conestat alfa, 2 reconstituted vials are needed
  Interventions: Drug: Conestat Alfa
- Placebo (Placebo Comparator): The comparator in the study will be a placebo, an isotonic sterile solution (pH 5.5 ± 0.3) for IV injection. The solution does not contain any preservatives. The placebo is formulated to match the study drug (conestat alfa) and is supplied in an identical single-dose IV bag. To maintain the blinding of the study, the IV bag containing the placebo will be indistinguishable from that containing conestat alfa, in addition to the labeling
  Interventions: Drug: Conestat Alfa

INTERVENTIONS:
Drug: Conestat Alfa — See arm/group descriptions
  Other Names: Ruconest

SUMMARY:
Angiotensin-converting enzyme inhibitors (ACE-Is), prescribed most often to treat hypertension, have been used extensively since the 1980s. Additional indications for their use include heart failure, diabetes mellitus, chronic kidney disease, and post-myocardial infarction. It is estimated that up to 40 million patients take ACE-Is worldwide. C1-INH is a serine protease inhibitor that is normally found in the blood. Its primary function is the regulation of the complement and contact system pathways by binding irreversibly to target proteases. It additionally inhibits the fibrinolytic, clotting, and kinin pathways.31 Patients with the hereditary forms of AE (HAE) tend to have lower quantitative or functional levels of C1-INH. This results in decreased suppression of plasma kallikrein and factor XIIa leading to cleavage of high molecular weight kininogen to form increased circulating levels of bradykinin. Bradykinin binds to bradykinin 2 receptors resulting in separation of endothelial vascular cells and extravasation of fluid manifesting clinically as angioedema. Conestat alfa (Ruconest®) is a recombinant human C1-INH that has been purified from the breast milk of genetically modified rabbits. It is a single-chain soluble glycoprotein that is made of 478 amino acids. Administering conestat alfa increases the amount of C1-INH in these patients, repleting their levels, and acting as a treatment for AE due to C1-INH deficiency. Conestat alfa has been studied on asymptomatic patients with HAE and was shown to dose-dependently increase the level of functional C1-INH. Additionally, it was shown to restore the level of the complement C4 protein, which is also decreased in these patients. Since the same pathophysiological pathway is involved in patients with ACE-I-induced AE, it is reasonable to hypothesize its effectiveness in the treatment of patients with acute attacks.

DETAILED DESCRIPTION:
This phase III clinical trial is being conducted to assess the benefits of emergency administration of intravenous (IV) conestat alfa to treat ACE-I-induced AE during an ED visit. This will be a multi-center, randomized, double-blind, two-armed, placebo-controlled trial. It will enroll 24 patients at two clinical sites in the United States. The population will consist of adult patients (≥ 18 years of age) who present to the ED with acute ACE-I-induced AE of the head and/or neck. Eligible patients will be enrolled in the study and randomized at a ratio of 1:1 to either the active treatment or placebo groups. The treatment group will receive intravenous conestat alfa at a fixed dose of 4200 International Units (IU) IV along with usual ED care at the discretion of the clinical care team, which may include epinephrine, H1 and/or H2-antihistamines, and corticosteroids. The placebo group will receive the same volume of an isotonic, sterile, normal saline (pH 5.5 ± 0.3) solution without any preservatives via IV injection, in addition to the usual care. Fixed dosing was chosen for this study rather than weight-based dosing as is used for treatment of acute attacks of hereditary angioedema because it is hypothesized that higher doses may have greater efficacy in ACE-I-induced AE and is safe to administer.32 A second fixed dose (4200 IU) of open label study drug will be administered 2 hours after the initial dose as a rescue medication if the subject has not experienced symptom relief (based upon TOSR evaluation). Additional doses of study drug or placebo will not be used. The rationale behind the dosage is based on the fact that 4200 IU is the maximum dose irrespective of patient weight. A second dose of the same amount is recommended if symptoms persist.

The primary objective is to compare the Time to Onset of Symptom Relief (TOSR) of conestat alfa compared to placebo in the treatment of ACE-I-induced AE. The secondary objective is to evaluate the efficacy of conestat alfa compared to placebo in Time to Meeting Discharge Criteria (TMDC), based on investigator-assessment of upper airway symptoms. The study will also compare the proportion of patients in each arm who 1) are hospitalized for any level of care 2) are admitted to the intensive care unit (ICU) and 3) requiring airway intervention (e.g., intubation, cricothyrotomy, or tracheotomy). Safety and tolerability of conestat alfa treatment will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older 2. Currently being treated with an ACE-I and presenting with presumed ACE-I-induced AE involving the head and/or neck region as determined by the clinical team 3. ACE-I-induced AE of the head and/or neck region of at least moderate severity within 24 hours of onset (must be sufficiently less than 24 hours to allow study drug to be administered within the same time frame) 4. AE that is at least moderate in severity for no less than one of the AE-associated airway symptoms (difficulty breathing, difficulty swallowing, voice changes, tongue swelling)32 5. Be able to provide informed consent or obtain informed consent from a legally appointed representative

-

Exclusion Criteria:

1. History of anaphylaxis, hypersensitivity, or allergic reactions to rabbits/rabbit-derived products and C1-INH preparations 2. Urticaria present during the current illness 3. AE thought by the clinical team to be due to any other etiology i.e., HAE (types I, II, and HAE with normal C1-INH), acquired AE, allergic/histaminergic AE 4. History of recent trauma, abscess, infection, local inflammation, local tumor, postoperative or post-radiogenic edema, salivary gland disorders, and non-ACE-I drug-induced AE 5. Family history of recurrent AE 6. History of AE prior to ACE-I therapy initiation 7. Last dose of ACE-I taken more than 72 hours before the onset of AE symptoms 8. History of a major systemic disease that is not well controlled (left to the study team's discretion) 9. Anyone requiring immediate airway intervention according to the clinical team, such as endotracheal intubation 10. Women who are pregnant or breast-feeding (pregnancy must be ruled out by a negative test with the exception of those who have undergone total hysterectomy, bilateral oophorectomy, or are 2 years post-menopausal) 11. Concurrent participation in other investigational drug studies 12. Treatment with other targeted therapeutic agents for HAE (ecallantide/icatibant/C1-INH/fresh frozen plasma) 13. In the opinion of the investigator, there is adequate response to the usual care treatments (epinephrine, H1 and/or H2 antihistamine, corticosteroids) within one hour before dosing of the study drug 14. Prisoners 15. Non-English speaking

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to assess the efficacy of conestat alfa compared to placebo in the treatment of ACE-1-induced AE based on the Time to Onset of Symptom Relief (TOSR) endpoint. | 24 hours
  The TOSR is defined as the time at which the total severity score of four airway compromising symptoms (difficulty breathing, difficulty swallowing, voice changes, and tongue swelling) has decreased by at least 1 point overall and no individual component of the score has increased. The 5-point severity scale is: 0 = absence of symptoms, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.

SECONDARY OUTCOMES:
The secondary objective is to compare the efficacy of conestat alfa to placebo for the treatment of ACE-1-induced AE based on the endpoint of Time to Meeting Discharge Criteria (TMDC). | 24 hours
  The criteria for discharge will be based on the assessment of the severity of four airway compromising symptoms, and will be calculated from the time of initiation of study drug administration to the earliest point at which the symptoms of difficulty breathing and difficulty swallowing have resolved (score = 0) and the symptoms of voice change and tongue swelling are mild or absent.

OTHER OUTCOMES:
Exploratory objective | 24 hours
  Exploratory objectives include comparison of the proportion of patients in each arm who 1) are hospitalized to any level of care 2) are admitted to the intensive care unit (ICU) and 3) required an airway intervention (e.g., intubation, cricothyrotomy, or tracheotomy).
Safety outcome | Every hour post treatment up to 8 hours and then every 2 hours from >8 to 24 hours; phone calls at day 7 and day 28.
  Safety and tolerability of conestat alfa treatment in patients experiencing ACE-I-induced AE will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Moellman, MD, Principal Investigator — University of Cincinnati; Gentry Wilkerson, MD, Principal Investigator — University of Maryland

IPD SHARING:
Plan to Share IPD: Yes
Data will be published. Raw data will be provided upon request as appropriate.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study will enrol over 12 months and data analysis and publication 0ver 6 to 12 months. Data will be available after publication of the study
Access Criteria: Contact the Protocol Chair Jonathan Bernstein or Co-PIs Drs. Joseph Moellman or Gentry Wilderson

REFERENCES:
- [Background] Bernstein JA, Moellman JJ, Collins SP, Hart KW, Lindsell CJ. Effectiveness of ecallantide in treating angiotensin-converting enzyme inhibitor-induced angioedema in the emergency department. Ann Allergy Asthma Immunol. 2015 Mar;114(3):245-9. doi: 10.1016/j.anai.2014.12.007. Epub 2015 Jan 16. PMID 25601538
- [Background] Moellman JJ, Bernstein JA, Lindsell C, Banerji A, Busse PJ, Camargo CA Jr, Collins SP, Craig TJ, Lumry WR, Nowak R, Pines JM, Raja AS, Riedl M, Ward MJ, Zuraw BL, Diercks D, Hiestand B, Campbell RL, Schneider S, Sinert R; American College of Allergy, Asthma & Immunology (ACAAI); Society for Academic Emergency Medicine (SAEM). A consensus parameter for the evaluation and management of angioedema in the emergency department. Acad Emerg Med. 2014 Apr;21(4):469-84. doi: 10.1111/acem.12341. PMID 24730413
- [Background] Bonner N, Panter C, Kimura A, Sinert R, Moellman J, Bernstein JA. Development and validation of the angiotensin-converting enzyme inhibitor (ACEI) induced angioedema investigator rating scale and proposed discharge criteria. BMC Health Serv Res. 2017 May 22;17(1):366. doi: 10.1186/s12913-017-2274-4. PMID 28532495
- [Background] Sinert R, Levy P, Bernstein JA, Body R, Sivilotti MLA, Moellman J, Schranz J, Baptista J, Kimura A, Nothaft W; CAMEO study group. Randomized Trial of Icatibant for Angiotensin-Converting Enzyme Inhibitor-Induced Upper Airway Angioedema. J Allergy Clin Immunol Pract. 2017 Sep-Oct;5(5):1402-1409.e3. doi: 10.1016/j.jaip.2017.03.003. Epub 2017 May 25. PMID 28552382
- [Background] Mudd PA, Hooker EA, Stolz U, Hart KW, Bernstein JA, Moellman JJ. Emergency department evaluation of patients with angiotensin converting enzyme inhibitor associated angioedema. Am J Emerg Med. 2020 Dec;38(12):2596-2601. doi: 10.1016/j.ajem.2019.12.058. Epub 2020 Jan 7. PMID 31932133
- [Background] Wilkerson RG, Dakessian A, Moellman JJ, Bernstein JA. Clinical trial of C1-INH for treatment of ACEi-induced angioedema. Am J Emerg Med. 2023 Jun;68:196-197. doi: 10.1016/j.ajem.2023.04.012. Epub 2023 Apr 11. No abstract available. PMID 37061431